CLINICAL TRIAL: NCT04052763
Title: Ability of FFR-CT to Detect the Absence of Hemodynamically Significant Lesions in Patients With High-risk Acute Coronary Syndrome Admitted in the Emergency Department With Chest Pain: a Diagnostic Accuracy Prospective Study
Brief Title: FFR-CT to Detect the Absence of Hemodynamically Significant Lesions in Patients With High-risk Acute Coronary Syndrome
Status: Terminated | Type: Observational
Why Stopped: Slow enrolment during the COVID pandemics
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr. Stephane Fournier, Chief Resident, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: no defined yet
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome
Keywords: NSTE-ACS; FFR-CT; FFRangio™
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- High-risk ACS patients: High-risk ACS patients admitted to the emergency departement witch chest pain.
  Interventions: Diagnostic Test: FFR-CT; Diagnostic Test: FFRangio™

INTERVENTIONS:
Diagnostic Test: FFR-CT — FFR-CT is a non invasive method using coronary CT images and 3 dimensional modelling to reconstruct coronary arteries and their stenoses, with subsequent calculation of fractional flow reserve (FFR) based on a mathematical algorithm.
Diagnostic Test: FFRangio™ — Angiography-derived FFR (FFRangio™) uses coronary angiography images and a mathematical algorithm to reconstruct a 3 dimensional model of coronary arteries with calculation of FFR without the use of a pressure guide.

SUMMARY:
The present study is a monocentric, observational, single arm, study, with the aim to determinate the ability of FFR-CT to exclude or confirm the presence of hemodynamically significant coronary stenosis, compared to coronary angiography in high-risk acute coronary syndrome patients.

DETAILED DESCRIPTION:
Study Design and Procedure:

The present study is a single arm, double blinded, prospective trial. Patients admitted to hospital with high-risk non-ST elevation acute coronary syndrome (NSTE-ACS) and who accept to participate to the study will undergo a coronary compute tomography (CT) angiography within 23 hours after diagnosis in order to have time to proceed to coronary angiography within the recommended window time of 24h. After realization of the CT, they will benefit from guidelines recommended treatment including a coronary angiography. According to internal and international guidelines, all efforts will be made to perform the coronary angiography within 24h of acute coronary syndrome (ACS) diagnosis.

The coronary CT angiography procedure takes approximately 1-2h (including logistical organization and patient transportation), and all efforts will be made not to delay the coronary angiography compared to patients who would not participate in the study. At the time of coronary angiography, patients will be blinded from the CT results as well as the direct treating physician and interventional cardiologist realizing the procedure, in order to avoid any influence in patients' management. The procedure will be done using a 256-slice multi-detector CT (GE Healthcare Revolution CT, Chicago, Illinois, USA). Just before the examination, as routinely done for this non-invasive test to allow for optimal coronary vasodilation and visualization, oral Metoprolol (25-50mg) will be administered if necessary to ensure a heart rate of 65 bpm or lower as well as one unique dose of sublingual nitroglycerine (400-800mg). Parameters used for CT acquisition will be as following: 100 Kilovoltage peak (kVp)/550 milliamperes (mA) for body mass index (BMI) <25 (high definition mode), 100 kVp/550 mA for BMI included between 25 and 30, 120 kVp/600 mA for BMI>30 (standard definition mode). Off line, an FFR-CT will be calculated with the data of the coronary CT angiography by blinded investigators in a central FFR-CT core laboratory (HeartFlow ®, Redwood City, CA 94063, USA). Hemodynamically significant lesion will be defined as lesion with an FFR-CT value of ≤ 0.80.

During the invasive coronary angiography, fractional flow reserve (FFR) will be measured in all lesions with a visual diameter stenosis ≥30% using the PressureWire™ X Guidewire (Abbott, Chicago, Illinois, USA) with the following protocol: first, equalization of the pressure wire and the aortic pressure will be performed at the tip of the guide catheter prior to all measurements. Second, the pressure wire will then be advanced distal to the stenosis. Third, hyperemia will be obtained using intracoronary adenosine (150mcg for the right coronary artery and 200mcg for the left descending or the circumflex coronary arteries). Fourth, at the end of the procedure, the absence of a drift will be confirmed after a pull-back of the pressure to the same location as the initial equalization. Hemodynamically significant lesion will be defined as lesion with an FFR value of ≤ 0.80.

Of note, in case of coronary angiography showing no obstructive coronary disease, and thus not offering satisfactory explanation for the myocardial injury, patients will undergo cardiac magnetic resonance imaging (CMRI), to detect a potential alternative diagnosis (myocarditis, Takotsubo…).

Both invasive FFR and FFR derived from FFR-CT will be compared with invasive FFR as gold standard.

Follow-up:

Follow-up will be organized 1 month (± 7 days), 6 months (± 14 days) and 12 months (± 14 days) after the acute coronary syndrome. These visits will include a detailed history, as well as physical examination and ECG. During the second visit, a transthoracic echocardiography will be performed, and a treadmill exercise stress test will be performed during the third visit.

Data and Statistical Analysis:

Statistical analysis will be carried out using SPSS 24.0 software (SPSS Inc., Chicago, Illinois) and Stata 14.3. Comparisons of characteristics of patients will be performed using Chi-squared tests for qualitative variables and Student's t or Mann-Whitney tests as appropriate. Confidence intervals (CI) for proportions (sensitivity, specificity, accuracy) will be calculated using the Wilson Score method. With the last iteration of the FFR-CT software, the per-patient sensitivity and specificity were 86% (95% CI: 77% to 92%) and 79% (95% CI: 72% to 84%). In the recent VERDICT trial based on NSTEMI patients, 12 % had 3 vessel disease, 23 % 2 vessel disease (which included left main), 34%, 1 vessel disease, 30% nothing, Thus, out of 100 patients with 300 coronaries, we expect 106 (i.e. 36+46+34) vessels with a stenosis. Based on the FAMOUS NSTEMI trial, 60% of invasive FFR measurements of these stenoses were significant. Thus, with a standard error of 0,05, and for a power of 80%, 204 patients will be required. However, some of the CT will not be suitable for analysis and some patients will have to be excluded. Therefore, we plan to include 250 patients. Of note, these number is also in line with the literature investigating the accuracy of FFR-CT versus FFR in patients with stable coronary artery disease.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years old patients
* Presenting a rise and/or fall of high-sensitive cardiac troponins T (hs-cTnt) values measured in Centre Hospitalier Universitaire Vaudois (CHUV) on at least 2 timepoints with at least one value above the 99th percentile of the upper range limit (URL) and with at least one of the following:
* Symptoms of ischemia
* New or presumed new significant ST-segment-T wave (ST-T) changes
* Informed consent signed
* Presumed availability for follow-up up to 1 year (i.e. patients only transiting through Switzerland for travel purpose are de facto excluded)
* Was transferred from CHUV Emergency Department to the CHUV Cardiology Service according to the fast-track institutional procedure

Exclusion criteria:

* STEMI patients
* Estimated glomerular filtration rate (eGFR) of <45 ml/min
* Presence of very high-risk criteria:
* Hemodynamic instability or cardiogenic shock
* Recurrent or ongoing chest pain refractory to medical treatment
* Life-threatening arrhythmias or cardiac arrest
* Mechanical complications of myocardial infarction
* Acute heart failure
* Recurrent dynamic ST-T wave changes, particularly with intermittent ST-elevation
* Pregnant and breast-feeding women (women of child bearing potential must have a negative urine or blood pregnancy at screening)
* Contra-indication to beta-blocker and/or nitroglycerin
* Patients transferred from another hospital where diagnosis was made using a troponin dosage other than hs-cTnT
* Patients with prior coronary artery bypass grafting (CABG)
* Patient with known severe heart failure (i.e Ejection fraction of left ventricle of <30%)
* Patient incapable of judgement or under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk acute coronary syndrome patients admitted to the emergency departement
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Negative predictive value of FFR-CT to detect the absence of hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Accuracy of FFR-CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Sensitivity of FFR-CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Specificity of FFR-CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Positive predictive value of FFR-CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high risk ACS patients | Through inclusion completion, expected after 18 months of enrolment

SECONDARY OUTCOMES:
Correlation (goodness of fit) of FFR-CT to detect hemodynamically significant stenosis, compared to invasive FFR in lesions with at least a 30% stenosis | Through inclusion completion, expected after 18 months of enrolment
Negative predictive value of coronary CT to detect the absence of hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Accuracy of coronary CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Sensibility of coronary CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Specificity of coronary CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Positive predictive value of coronary CT to detect hemodynamically significant stenosis, compared to angiography (with FFR in case of lesion with at least a 30% stenosis) in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Safety endpoint | Through inclusion completion, expected after 18 months of enrolment
  Composite endpoint composed of: radiation dose received per patient, dose of iodinated contrast media received per patient, incidence of acute kidney failure defined as an increase of > 1.5x the baseline creatinine value 3 days after the coronary angiography, incidence of vascular complications related to the coronary angiogram, incidence of stroke, and incidence of MACEs (major adverse cardiac events)
Feasibility of an FFR-CT strategy in case of high-risk ACS, defined as the number of cases among enrolled patients where CT and FFR-CT is not feasible (moving artefacts, quality…) | Through inclusion completion, expected after 18 months of enrolment
Accuracy, of FFRangio™ to detect hemodynamically significant stenosis, as compared to invasive FFR in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Sensitivity of FFRangio™ to detect hemodynamically significant stenosis, as compared to invasive FFR in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Specificity of FFRangio™ to detect hemodynamically significant stenosis, as compared to invasive FFR in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Negative predictive value of FFRangio™ to detect hemodynamically significant stenosis, as compared to invasive FFR in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Positive predictive value of FFRangio™ to detect hemodynamically significant stenosis, as compared to invasive FFR in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Accuracy of FFRangio™ to detect hemodynamically significant stenosis, compared to FFR-CT in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Sensitivity of FFRangio™ to detect hemodynamically significant stenosis, compared to FFR-CT in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Specificity of FFRangio™ to detect hemodynamically significant stenosis, compared to FFR-CT in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Negative predictive value of FFRangio™ to detect hemodynamically significant stenosis, compared to FFR-CT in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Positive predictive value of FFRangio™ to detect hemodynamically significant stenosis, compared to FFR-CT in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Distribution of treatment assignement (PCI, CABG, medical treatment), based on angiography versus treatment decision according to invasive FFR in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Distribution of treatment assignement (PCI, CABG, medical treatment), based on angiography versus treatment decision according to FFRangio™ in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Distribution of treatment assignement (PCI, CABG, medical treatment), based on angiography versus treatment decision according to FFR-CT in high-risk ACS patients | Through inclusion completion, expected after 18 months of enrolment
Natural history of deferred lesions according to invasive FFR in term of major adverse cardiac events (MACE) | Through follow-up completion, expected 30 months after study initiation
Natural history of deferred lesions according to FFR-CT, in term of major adverse cardiac events (MACE) | Through follow-up completion, expected 30 months after study initiation
Natural history of deferred lesions according to CT in term of major adverse cardiac events (MACE) | Through follow-up completion, expected 30 months after study initiation
Natural history of deferred lesions according to FFRangio™ in term of major adverse cardiac events (MACE) | Through follow-up completion, expected 30 months after study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Fournier, MD, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland